CLINICAL TRIAL: NCT00954187
Title: Comparison of Oral Gabapentin and Pregabalin in Postoperative Pain Control After Photorefractive Keratectomy: a Prospective, Randomized Study.
Brief Title: Comparison of Oral Gabapentin and Pregabalin in Postoperative Pain Control After Photorefractive Keratectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 59070
Record Dates: First submitted 2009-08-05; First posted 2009-08-07 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Gabapentin; Pregabalin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gabapentin (Experimental): Neurontin
  Interventions: Drug: Gabapentin
- Pregabalin (Experimental): Lyrica
  Interventions: Drug: pregabalin

INTERVENTIONS:
Drug: Gabapentin — Gabapentin - 300 mg three times a day starting two hours prior to surgery and will continue for a total of four days
  Other Names: Neurontin
  Arms: Gabapentin
Drug: pregabalin — 50 mg PO TID
  Other Names: Lyrica
  Arms: Pregabalin

SUMMARY:
Purpose: To compare the efficacy of oral gabapentin and its newer analogue pregabalin in postoperative pain control after photorefractive keratectomy (PRK).

Methods: One hundred and four patients who meet the inclusion criteria undergoing PRK in one or both eyes will be randomized into one of two treatment groups. Those in group A will be treated with gabapentin, and those in group B will be treated with pregabalin to control postoperative PRK pain. Patients in both groups will begin treatment two hours prior to surgery in order to achieve therapeutic blood levels of each medication. After surgery the patients will assess their pain level using the visual analogue scale (VAS) at different intervals of time - one hour after surgery, the evening of the surgery, and three times each day for three subsequent days. Patients will also daily assess their level of somnolence using the Epworth Sleepiness Scale (ESS) and record the presence of dizziness for the same amount of time. On the fourth day they will return to clinic for a postoperative appointment. At that time the pain, sleepiness, and dizziness assessment scales will be collected and analyzed. The patients will return one month later to further assess long-term pain and healing after PRK.

Results: Both gabapentin and pregabalin have been shown in previous studies to treat postoperative pain effectively. The effects of gabapentin 300 mg TID for 3 days versus pregabalin 50 mg TID for 3 days on decreasing overall postoperative pain following PRK will be presented.

Conclusion: The effectiveness of the two different treatment medications will be analyzed, and the conclusion will be based on the results.

DETAILED DESCRIPTION:
METHODS:

One hundred and four patients who meet the inclusion criteria undergoing photorefractive keratectomy (PRK) in one or both eyes will be randomly assigned into one of two treatment groups via computer. Those in group A will be treated with gabapentin and those in group B will be treated with pregabalin to control postoperative PRK pain. Patients in both groups will begin treatment two hours prior to surgery. Patients in the gabapentin group will take 300 mg three times a day starting two hours prior to surgery and will continue for a total of four days. Patients in the pregabalin group will take 50 mg three times a day starting two hours prior to surgery and will also continue for four days.

Only the refractive surgery coordinator and the patient will know what medication the patient is taking. The patient will be instructed not to share this information with any other study participants or their surgeon. The coordinator will keep a list of the patients ID numbers and the treatments they are receiving.

Prior to surgery, each patient will be taught how to assess their pain level using the visual analogue scale (VAS), a well documented method of pain assessment. After surgery the patients will assess their pain levels at different intervals of time - one hour after surgery, the evening of the surgery, and three times a day for four subsequent days. Patients will also daily assess their level of somnolence using the Epworth Sleepiness Scale (ESS) and record the presence of dizziness daily for the same amount of time. On the fourth day they will return to clinic for a post operative appointment. At that time the pain assessment scales will be collected and analyzed. The patients will return at one month to further assess long term pain after PRK.

Statistical Analysis:

Postoperative pain levels recorded using the visual analogue scales, ESS, and self reported dizziness assessments will be collected on the fourth postoperative day. These will be compiled into data sets and analyzed. Data will be compiled into means with lower and upper quartiles and analyzed using a two-sided t test. The difference in pain levels will be described throughout the postoperative period to determine if one medication significantly reduces postoperative pain initially within the first 24 hours, during the interval between 24 hours to four days, and further after surgery (one month postoperatively). Data regarding levels of somnolence and dizziness will also be reported.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Undergoing PRK in at least one eye

Exclusion Criteria:

* Serious medical problems within the last 6 months including myocardial infarction (heart attack), congestive heart failure, stroke, deep vein thrombosis, pulmonary embolism, and other conditions, etc.
* Serious kidney disease as evidenced by the need for dialysis or kidney transplant.
* History of seizure or other neurologic disorders.
* Patients intending to become pregnant or who are pregnant or nursing over the projected course of treatment.
* Currently taking gabapentin or pregabalin for other medical purposes.
* Known allergic reaction to gabapentin or pregabalin from previous use.
* Plans to move out of the area within 8 weeks after the surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-11; Primary Completion 2012-09 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julio Narvaez, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University - Ophthalmology, Loma Linda, California, United States

REFERENCES:
- [Background] Shortt AJ, Allan BD. Photorefractive keratectomy (PRK) versus laser-assisted in-situ keratomileusis (LASIK) for myopia. Cochrane Database Syst Rev. 2006 Apr 19;(2):CD005135. doi: 10.1002/14651858.CD005135.pub2. PMID 16625626
- [Background] Ambrosio R Jr, Wilson S. LASIK vs LASEK vs PRK: advantages and indications. Semin Ophthalmol. 2003 Mar;18(1):2-10. doi: 10.1076/soph.18.1.2.14074. PMID 12759854
- [Background] Lee JB, Kim JS, Choe C, Seong GJ, Kim EK. Comparison of two procedures: photorefractive keratectomy versus laser in situ keratomileusis for low to moderate myopia. Jpn J Ophthalmol. 2001 Sep-Oct;45(5):487-91. doi: 10.1016/s0021-5155(01)00406-3. PMID 11583670
- [Background] Van de Pol C, Greig JL, Estrada A, Bissette GM, Bower KS. Visual and flight performance recovery after PRK or LASIK in helicopter pilots. Aviat Space Environ Med. 2007 Jun;78(6):547-53. PMID 17571652
- [Background] Walker MB, Wilson SE. Recovery of uncorrected visual acuity after laser in situ keratomileusis or photorefractive keratectomy for low myopia. Cornea. 2001 Mar;20(2):153-5. doi: 10.1097/00003226-200103000-00007. PMID 11248818
- [Background] Sandoval HP, de Castro LE, Vroman DT, Solomon KD. Refractive Surgery Survey 2004. J Cataract Refract Surg. 2005 Jan;31(1):221-33. doi: 10.1016/j.jcrs.2004.08.047. PMID 15721716
- [Background] Hazelrigg SR, Auer JE, Seifert PE. Experience in 100 transthoracic balloon pumps. Ann Thorac Surg. 1992 Sep;54(3):528-32. doi: 10.1016/0003-4975(92)90448-d. PMID 1510521
- [Background] Dirks J, Fredensborg BB, Christensen D, Fomsgaard JS, Flyger H, Dahl JB. A randomized study of the effects of single-dose gabapentin versus placebo on postoperative pain and morphine consumption after mastectomy. Anesthesiology. 2002 Sep;97(3):560-4. doi: 10.1097/00000542-200209000-00007. PMID 12218520
- [Background] Fassoulaki A, Patris K, Sarantopoulos C, Hogan Q. The analgesic effect of gabapentin and mexiletine after breast surgery for cancer. Anesth Analg. 2002 Oct;95(4):985-91, table of contents. doi: 10.1097/00000539-200210000-00036. PMID 12351281
- [Background] Pandey CK, Navkar DV, Giri PJ, Raza M, Behari S, Singh RB, Singh U, Singh PK. Evaluation of the optimal preemptive dose of gabapentin for postoperative pain relief after lumbar diskectomy: a randomized, double-blind, placebo-controlled study. J Neurosurg Anesthesiol. 2005 Apr;17(2):65-8. doi: 10.1097/01.ana.0000151407.62650.51. PMID 15840990
- [Background] Turan A, Karamanlioglu B, Memis D, Hamamcioglu MK, Tukenmez B, Pamukcu Z, Kurt I. Analgesic effects of gabapentin after spinal surgery. Anesthesiology. 2004 Apr;100(4):935-8. doi: 10.1097/00000542-200404000-00025. PMID 15087630
- [Background] Turan A, Memis D, Karamanlioglu B, Yagiz R, Pamukcu Z, Yavuz E. The analgesic effects of gabapentin in monitored anesthesia care for ear-nose-throat surgery. Anesth Analg. 2004 Aug;99(2):375-8, table of contents. doi: 10.1213/01.ANE.0000136646.11737.7B. PMID 15271709
- [Background] Menigaux C, Adam F, Guignard B, Sessler DI, Chauvin M. Preoperative gabapentin decreases anxiety and improves early functional recovery from knee surgery. Anesth Analg. 2005 May;100(5):1394-1399. doi: 10.1213/01.ANE.0000152010.74739.B8. PMID 15845693
- [Background] Kavalieratos CS, Dimou T. Gabapentin therapy for painful, blind glaucomatous eye: case report. Pain Med. 2008 Apr;9(3):377-8. doi: 10.1111/j.1526-4637.2006.00167.x. PMID 18366517
- [Background] Poujois A, Vidailhet M, Trocello JM, Bourdain F, Gaymard B, Rivaud-Pechoux S. Effect of gabapentin on oculomotor control and parkinsonism in patients with progressive supranuclear palsy. Eur J Neurol. 2007 Sep;14(9):1060-2. doi: 10.1111/j.1468-1331.2007.01687.x. PMID 17718702
- [Background] Rahman W, Proudlock F, Gottlob I. Oral gabapentin treatment for symptomatic Heimann-Bielschowsky phenomenon. Am J Ophthalmol. 2006 Jan;141(1):221-2. doi: 10.1016/j.ajo.2005.08.022. PMID 16387013
- [Background] Choudhuri I, Sarvananthan N, Gottlob I. Survey of management of acquired nystagmus in the United Kingdom. Eye (Lond). 2007 Sep;21(9):1194-7. doi: 10.1038/sj.eye.6702434. Epub 2006 May 26. PMID 16732211
- [Background] Nissman SA, Tractenberg RE, Babbar-Goel A, Pasternak JF. Oral gabapentin for the treatment of postoperative pain after photorefractive keratectomy. Am J Ophthalmol. 2008 Apr;145(4):623-629. doi: 10.1016/j.ajo.2007.11.012. Epub 2008 Jan 28. PMID 18226799
- [Background] Agarwal A, Gautam S, Gupta D, Agarwal S, Singh PK, Singh U. Evaluation of a single preoperative dose of pregabalin for attenuation of postoperative pain after laparoscopic cholecystectomy. Br J Anaesth. 2008 Nov;101(5):700-4. doi: 10.1093/bja/aen244. Epub 2008 Aug 20. PMID 18716003
- [Background] Taylor CP. Mechanisms of analgesia by gabapentin and pregabalin--calcium channel alpha2-delta [Cavalpha2-delta] ligands. Pain. 2009 Mar;142(1-2):13-6. doi: 10.1016/j.pain.2008.11.019. Epub 2009 Jan 6. No abstract available. PMID 19128880
- [Background] Guay DR. Pregabalin in neuropathic pain: a more "pharmaceutically elegant" gabapentin? Am J Geriatr Pharmacother. 2005 Dec;3(4):274-87. PMID 16503325
- [Background] Lesser H, Sharma U, LaMoreaux L, Poole RM. Pregabalin relieves symptoms of painful diabetic neuropathy: a randomized controlled trial. Neurology. 2004 Dec 14;63(11):2104-10. doi: 10.1212/01.wnl.0000145767.36287.a1. PMID 15596757
- [Background] Richter RW, Portenoy R, Sharma U, Lamoreaux L, Bockbrader H, Knapp LE. Relief of painful diabetic peripheral neuropathy with pregabalin: a randomized, placebo-controlled trial. J Pain. 2005 Apr;6(4):253-60. doi: 10.1016/j.jpain.2004.12.007. PMID 15820913
- [Background] Huskisson EC. Measurement of pain. Lancet. 1974 Nov 9;2(7889):1127-31. doi: 10.1016/s0140-6736(74)90884-8. No abstract available. PMID 4139420
- [Background] Scott J, Huskisson EC. Graphic representation of pain. Pain. 1976 Jun;2(2):175-84. No abstract available. PMID 1026900
- [Background] Revill SI, Robinson JO, Rosen M, Hogg MI. The reliability of a linear analogue for evaluating pain. Anaesthesia. 1976 Nov;31(9):1191-8. doi: 10.1111/j.1365-2044.1976.tb11971.x. PMID 1015603

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gabapentin | Pregabalin
Started | 0 (No subjects were assigned treatment and no study procedures were performed) | 0 (No subjects were assigned treatment and no study procedures were performed)
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No subjects were randomized and assigned treatment so Baseline Characteristics were not collected
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin | Pregabalin | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous
Gender
  Female |  |  | 0
  Male |  |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Decreased Overall Pain Score as Measured by the Visual Analogue Scale
Description: No data was collected or analyzed. No study procedures were performed.
Time Frame: one month
Population: No subjects were assigned treatment and no study procedures were performed
Arm/Group | Gabapentin | Pregabalin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Gabapentin | Pregabalin
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes